CLINICAL TRIAL: NCT04165707
Title: A Randomized Controlled Trial Comparing Weight Loss Effects Between the Keyto Virtual "Ketogenic Diet" Program Compared to a Standard-care Weight Loss App
Brief Title: A Weight Loss RCT Comparing Keyto vs Weight Watchers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H19-01341
Record Dates: First submitted 2019-11-06; First posted 2019-11-18 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Overweight and Obesity; Ketogenic Diet
Keywords: diet; weight loss; ketogenic diet; low carbohydrate
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Keyto intervention arm (Experimental): Keyto device + app
  Interventions: Device: Keyto device + app
- Weight Watchers comparator arm (Active Comparator): Weight Watchers app
  Interventions: Other: Weight Watchers app

INTERVENTIONS:
Device: Keyto device + app — Keyto is a self-monitoring and app-enhanced intervention to help individuals learn about and monitor their breath acetone (a measure of ketosis) levels to promote a very low carbohydrate diet and weight loss.
  Arms: Keyto intervention arm
Other: Weight Watchers app — The Weight Watchers app helps people to monitor their food intake, track points and provides recipe ideas to support weight loss.
  Arms: Weight Watchers comparator arm

SUMMARY:
Very low-carbohydrate ketogenic diet may have beneficial metabolic and weight loss effects, however, adhering to this diet may be challenging. Keyto is a self-monitoring and app-enhanced intervention to help individuals learn about and monitor their breath acetone (a measure of ketosis) levels to promote dietary change and weight loss. The purpose of this research is to test the Keyto self-monitoring + app intervention against a "standard of care" weight loss dietary app (Weight Watchers). 144 participants will be recruited through Facebook ads, provide online consent, and will be randomized to one of the two conditions. Weight loss after 12 weeks will be assessed as the primary outcome, with weight loss at 24 and 48 weeks being secondary outcomes. Blood samples will be collected at baseline and 12 weeks with optional blood samples at 48 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Living in the State of California
* Body mass index (BMI) 27-43
* Must speak, read, and comprehend English
* Access to reliable internet and wi-fi
* Must have a valid email address and phone number
* Must have an Apple iPhone (iPhone 7 or later, iOS 11 or later) with cellular data plan
* Must have a kitchen and be willing to cook
* Willingness to reduce carbohydrate intake to less than 30g/day
* Willingness to restrict intake of added sugar, bread, grain, rice, pasta, sweets, most fruits, pastries, and other carbohydrates
* Willingness to comply with a strict diet for 12 months
* Willingness to eat a diet that is primarily plant and fish-based
* Interest in losing weight

Exclusion Criteria:

* HIV or immunocompromised
* Current or past cancer diagnosis
* Pregnant, breastfeeding, or planned pregnancy in next 12 months
* Beginning or ending hormonal contraception in next 12 months
* Current diagnosis of diabetes
* History of heart attack or stent
* Currently taking glucose-lowering drugs, statins, or oral steroids
* History of gastric bypass surgery or any other weight-loss surgery
* History of anorexia or bulimia
* History of mental illness
* Current smoker or smoked cigarettes within past 12 months
* Currently eating fewer than 50 g carbohydrates per day
* Have tried a low-carb, high fat (ketogenic diet) within the past 3 months
* Recent weight loss or gain of more than 5% body weight in past 6 months
* Previous experience with the Weight Watchers diet app
* Experience with a low-carbohydrate of ketogenic diet within past 6 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Change in body mass at 12 weeks | 12 weeks from baseline
  Change in body mass (in kilograms)

SECONDARY OUTCOMES:
Change in body mass at 24 and 48 weeks | 24 and 48 weeks from baseline
  Change in body mass (in kilograms)
Carbohydrate intake | 12, 24, and 48 weeks from baseline
  Total consumption of carbohydrates in 24 hour period (in grams)
Total fat intake | 12, 24, and 48 weeks from baseline
  Total consumption of fat in 24 hour period (in grams)
Saturated fat intake | 12, 24, and 48 weeks from baseline
  Total consumption of saturated fat in 24 hour period (in grams)
Polyunsaturated fat intake | 12, 24, and 48 weeks from baseline
  Total consumption of polyunsaturated fat in 24 hour period (in grams)
Monounsaturated fat intake | 12, 24, and 48 weeks from baseline
  Total consumption of monounsaturated fat in 24 hour period (in grams)
Total energy intake | 12, 24, and 48 weeks from baseline
  Total energy intake in 24 hour period (in kilocalories)
HbA1C | 12 and 48 weeks from baseline
  Blood test will be used to determine changes in HbA1C
Fasting glucose | 12 and 48 weeks from baseline
  Blood test will be used to determine changes in fasting serum glucose
Fasting insulin | 12 and 48 weeks from baseline
  Blood test will be used to determine changes in fasting serum insulin
Fasting high-sensitivity C-reactive protein | 12 and 48 weeks from baseline
  Blood test will be used to determine changes in fasting serum high-sensitivity C-reactive protein
Fasting homeostasis model assessment of insulin resistance (HOMA-IR) | 12 and 48 weeks from baseline
  Blood test will be used to determine changes in HOMA-IR
Fasting total cholesterol | 12 and 48 weeks from baseline
  Blood test will be used to determine changes in serum total cholesterol
Fasting high-density lipoprotein (HDL) cholesterol | 12 and 48 weeks from baseline
  Blood test will be used to determine changes in serum HDL cholesterol
Fasting lipoprotein fractions | 12 and 48 weeks from baseline
  Blood test will determine changes in serum lipoprotein fractions measured by ion mobility
Fasting lipoprotein (a) | 12 and 48 weeks from baseline
  Blood test will determine changes in serum lipoprotein (a)
Fasting triglycerides | 12 and 48 weeks from baseline
  Blood test will determine changes in serum trigylcerides
Fasting non-HDL cholesterol | 12 and 48 weeks from baseline
  Blood test will determine changes in serum non-HDL cholesterol

OTHER OUTCOMES:
Fasting albumin | 12 and 48 weeks from baseline
  Blood test will determine changes in serum albumin
Fasting globulin | 12 and 48 weeks from baseline
  Blood test will determine changes in serum globulin
Fasting total bilirubin | 12 and 48 weeks from baseline
  Blood test will determine changes in serum bilirubin
Fasting alkaline phosphatase | 12 and 48 weeks from baseline
  Blood test will determine changes in serum alkaline phosphatase
Fasting aspartate aminotransferase | 12 and 48 weeks from baseline
  Blood test will determine changes in serum aspartate aminotransferase
Fasting alanine aminotransferase | 12 and 48 weeks from baseline
  Blood test will determine changes in serum alanine aminotransferase

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Little, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

REFERENCES:
- [Derived] Falkenhain K, Lowe DA, Locke SR, Singer J, Weiss EJ, Little JP. Long-Term Weight Loss in Adults With Overweight or Obesity Using a Breath Biofeedback mHealth App: A One-Year Follow-Up of a Randomized Trial. Obes Sci Pract. 2025 Dec 5;11(6):e70106. doi: 10.1002/osp4.70106. eCollection 2025 Dec. PMID 41356752
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Falkenhain K, Locke SR, Lowe DA, Lee T, Singer J, Weiss EJ, Little JP. Use of an mHealth Ketogenic Diet App Intervention and User Behaviors Associated With Weight Loss in Adults With Overweight or Obesity: Secondary Analysis of a Randomized Clinical Trial. JMIR Mhealth Uhealth. 2022 Mar 14;10(3):e33940. doi: 10.2196/33940. PMID 35285809
- [Derived] Locke SR, Falkenhain K, Lowe DA, Lee T, Singer J, Weiss EJ, Little JP. Comparing the Keyto App and Device with Weight Watchers' WW App for Weight Loss: Protocol for a Randomized Trial. JMIR Res Protoc. 2020 Aug 17;9(8):e19053. doi: 10.2196/19053. PMID 32804087